CLINICAL TRIAL: NCT00493857
Title: A Phase II Open-Label, 2-Cohort Study of Nimotuzumab 400 mg Weekly Plus Irinotecan (Cohort 1) and Nimotuzumab 400 mg Every 2 Weeks Plus Irinotecan (Cohort 2) in Patients With Irinotecan-Refractory Metastatic Colorectal Cancer
Brief Title: Study of Nimotuzumab and Irinotecan in Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Cohort 2 not going forward. Manadate changes in Company
Sponsor: YM BioSciences (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YMB 1000-015
Record Dates: First submitted 2007-06-27; First posted 2007-06-28 (Estimated); Last update posted 2008-11-17 (Estimated); Status verified 2008-11

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; Monoclonal antibody; Anti-EGFR
MeSH Terms: conditions — Colorectal Neoplasms | interventions — nimotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 2 (Experimental): Nimotuzumab 400mg every week or every two weeks
  Interventions: Drug: Nimotuzumab Humanized Monoclonal Antibody; Drug: Nimotuzumab

INTERVENTIONS:
Drug: Nimotuzumab Humanized Monoclonal Antibody — Nimotuzumab 400mg every week
Drug: Nimotuzumab — Nimotuzumab 400mg every 2 weeks

SUMMARY:
This study will determine if nimotuzumab provides a benefit in this type of cancer when given in combination with irinotecan.

The study will test:

* How long any good effects last.
* How bad any side effects are.

Objectives:

Primary:

The primary goal is to assess the Objective Response Rate (ORR) that the combination of irinotecan and nimotuzumab will produce in patients with irinotecan-refractory metastatic colorectal cancer

Secondary:

* To assess the incidence of Grade 2 or greater acneiform rash or infusion reaction, allergic reaction or anaphylactoid reaction AEs in patients with irinotecan-refractory metastatic colorectal cancer following weekly or 2-weekly nimotuzumab schedules;
* To assess Progression-Free Survival (PFS), defined as time from date of randomization until date of disease progression (clinical or radiological) or death due to any cause, for the two nimotuzumab schedules;
* To assess the rates and durations of Stable Disease (SD) following weekly or 2-weekly nimotuzumab schedules;
* To assess the Time to Disease Progression (TTP) following weekly or 2-weekly nimotuzumab schedules;
* To evaluate ORR in patients who are identified as having "primary" irinotecan resistance following weekly or 2-weekly nimotuzumab schedules;
* To evaluate Overall Survival (OS) following weekly or 2-weekly nimotuzumab schedules;
* To compare the two dosing schedules of nimotuzumab with respect to objective response rates and safety;
* To evaluate the overall safety and toxicity profiles of these two dose regimens of nimotuzumab;
* To evaluate trough levels and accumulation of nimotuzumab in serum of patients receiving the drug on weekly or 2-weekly regimens.

DETAILED DESCRIPTION:
The patient will receive nimotuzumab every 2 weeks plus irinotecan. Nimotuzumab will be given at a dose of 400 mg once every 2 weeks for 12 weeks. Irinotecan will be given at the same dose and schedule as the last dose and schedule given during the most recent pre-study irinotecan containing therapy. If the tumour does not show signs of further growth after 12 weeks of treatment, the patient will continue receiving nimotuzumab 400 mg every 2 weeks for up to 18 months or as long as they are getting a benefit from the drug.

ELIGIBILITY:
Inclusion Criteria

* Confirmed colorectal cancer with metastatic disease documented on diagnostic imaging studies.
* Measurable disease,
* Must have clinical documentation of failure after receiving at least one chemotherapy regimen for metastatic disease that contained irinotecan.
* Must have documentation of failure by CT, MRI or PET scan. Patients who were intolerant of irinotecan despite dose attenuations are not eligible for this trial.
* Patients must have failed irinotecan which they received on one of the following three starting regimens:Weekly,Biweekly or every 3 weeks. mg/m2.

  6.Patients may have received any number of prior standard and investigational regimens or radiation treatments, provided that they meet all other eligibility criteria.
* Age greater than 18 years.
* Life expectancy of greater than 3 months.
* ECOG performance status less than 1
* Patients must have normal organ and marrow function
* Patients must have medical documentation of dose, schedule, and dates of last irinotecan administration.
* Women of child-bearing potential and men must agree to use adequate contraception
* Patients must have the ability to understand and the willingness to sign a written informed consent document.

Subject Exclusion Criteria

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier. Neurotoxicity, if present, must have recovered to < grade 2.
* No other investigational agents.
* No known brain metastases.Patients with a history of primary CNS tumours, seizures not well controlled with standard medical therapy, or history of stroke will also be excluded.
* History of allergic reactions attributed to compounds of chemical or biologic composition similar to nimotuzumab, irinotecan, or other agents used in the study.
* Previous EGFR-directed therapy
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring parenteral antibiotics, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled hypertension, clinically significant cardiac arrhythmia, history of myocardial infarction within the past 6 months, or psychiatric illness/social situations that would limit compliance with study requirements.
* HIV-positive patients on combination antiretroviral therapy are ineligible
* Active cardiovascular disease, e.g., uncontrolled hypertension, unstable angina, New York Heart Association grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medications, or grade II or greater peripheral vascular disease. In addition, patients with arterial thrombosis, myocardial infarction, and cerebral vascular accidents [stroke/transient ischemic attack (TIA)] within 6 months prior to study entry will be excluded.
* Organ allografts requiring immunosuppressive therapy. -.Pregnant or lactating women are excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-06; Primary Completion 2008-08 (Actual); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
The primary goal is to assess the Objective Response Rate (ORR) that the combination of irinotecan and nimotuzumab will produce in patients with irinotecan-refractory metastatic colorectal cancer | 18-24 months

SECONDARY OUTCOMES:
Assess the incidence of acneiform rash,drug reaction,adverse events, the assessment of progression-free survival,stable disease,time to disease progression, overall survival, objective response rates, safety and trough levels in the serum of patients. | 18-24 months

CONTACTS AND LOCATIONS:
Overall Officials: Amil Shah, MD, Study Chair — Vancouver Cancer Centre BC cancer Agency
Locations (12):
- Canada (12):
  - Tom Baker Cancer Center, Calgary, Alberta
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - Dr. H. Bliss Purphy Cancer Centre, St. John's, Newfoundland and Labrador
  - Royal Victoria Hospital, Barrie, Ontario
  - Grand River Hospital, Kitchener, Ontario
  - London Regional Cancer Centre, London, Ontario
  - Credit Valley Hospital /Carlo Fidani Peel Regional Cancer Centre, Mississauga, Ontario
  - Cancer Care Program Southlake Regional Health Centre, Newmarket, Ontario
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Algoma District Cancer Care Program, Sault Ste. Marie, Ontario
  - Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario